CLINICAL TRIAL: NCT01593098
Title: A Prospective Study Into the Risk of Colorectal Neoplasms in Individuals With a Family History of Advanced Adenomas (Sibling AN Study)
Acronym: AN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor of Medicine, Chinese University of Hong Kong
Other Study IDs: AN study
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Adenoma; CRC
Keywords: siblings; advanced neoplasm; mRNA; TaqMan microRNA expression assays
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colonic biopsies, blood, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed siblings: Siblings (age >40 and <70) of individuals diagnosed with advanced neoplasm on screening colonoscopy. Advanced neoplasm is defined as adenomas≥10mm size, >25% villous features, severe dysplasia or carcinoma-in-situ
- unexposed siblings: Siblings (age >40 and <70) of individuals diagnosed with no polyp on screening colonoscopy who is age and sex matched to case.

SUMMARY:
To prospectively determine the prevalence of colorectal neoplasia in siblings of Hong Kong Chinese patients with advanced neoplasm compared with a sex and age-matched control population. To determine the molecular alteration profiles of colonic adenomas in siblings of patients with advanced neoplasm

DETAILED DESCRIPTION:
The incidence of colorectal cancer (CRC) is rising rapidly in Hong Kong. It is the second commonest cancer in Hong Kong with more than 4000 new cases diagnosed in 2007, and it is also the second commonest cause of cancer death accounting for approximately 1,700 deaths per year. It has been estimated that 1 in 20 (5%) and 1 in 33 (3%) Hong Kong males and females, respectively, will develop CRC in their life time. (1) Data from the Hong Kong cancer registry showed that almost half of the cancer cases were stage III or IV disease at diagnosis which was associated with a worse prognosis(1), suggesting that earlier detection of CRC is important.

Genetic factors play an important role in the development of CRC. Approximately one fifth of CRC are associated with familial clustering(2), whilst hereditary syndromes including hereditary non- polyposis colorectal cancer (HNPCC) and familial adenomatous polyposis (FAP) account for approximately six percent of CRC cases (3;4)

Individuals with a family history of CRC have an increased risk of developing colonic neoplasm (cancer and adenoma). Meta-analyses of epidemiological studies showed that FDR of patients with CRC have an approximately two to three-fold increase risk of developing CRC compared with the general population (5-9). [Table 1]. The frequency of adenomas (12-69%) is also higher in relatives of patients with CRC although most of the earlier data have been derived from cohort studies (10-16). In the recent two case-control studies, the choice of the control population has been questionable (17;18) [Table 2]. Our own case-control study of screening colonoscopy in FDR with CRC, compared with FDR of patients with a normal colonoscopy ( published in abstract form) showed that the prevalence of colonic adenomas was significantly higher in cases compared with controls (25.3% versus 15.6%) (19).

Colorectal adenomas are precursors of CRC, and FDR of individuals with colonic adenomas also have an increased risk of CRC as well as colonic adenomas (20;21) The risk of developing colorectal neoplasia in FDR of patients with adenoma is likely be influenced by the characteristics of the adenoma in the index case. Colonic adenomas have a higher malignancy potential when they are greater than 10mm in size, and / or contains a villous component or severe dysplasia (22). In one study, relative risk of CRC for FDR was higher in relatives of patients with large adenomas (>10mm) than in those with small adenomas (OR 2.1 and 1.2 respectively) (23). These findings have been reproduced in a recent study from France, which in addition showed that the risk was particularly high if the index case was younger than 60 years at diagnosis of a large adenoma, male or if they had a large adenoma in the left colon (24). In a separate study, relatives of patients with advanced neoplasm (OR1.62), but not those with small tubular adenomas (OR 1.26), have an increased risk of CRC (25).

Little is known about the prevalence of CRC and adenomas among siblings of individuals with advanced neoplasm in Hong Kong. Furthermore screening procedure for relatives of patients with high risk adenomas are not as well established as screening strategies for relatives of patients with CRC. This information is of important relevance in the formulation of an effective CRC screening strategy in Hong Kong (26). In a pilot screening project in 2001 among asymptomatic subjects of greater than 50 years old, the investigator have demonstrated an approximately 12% rate of advanced neoplasms using colonoscopy as a tool. Since 2008, asymptomatic subjects greater than 50 years old have been invited to undergo colonoscopy screening for CRC in PWH and AHNH hospital. To date about 1800 asymptomatic subjects have completed colonoscopy screening. This project provides the investigators with the opportunity to use an original design to determine the prevalence of colorectal neoplasia in siblings of patients with advanced neoplasm, compared with siblings of asymptomatic individuals who have had a negative screening colonoscopy during the same period of time.

The molecular pathways leading to tumour development in familial colorectal neoplasms are likely to be different from sporadic cases. Development of new molecular based methods for early detection, prevention or treatment relies heavily on the understanding of the differences between sporadic and familial neoplasms. Identification of genetic mutations can also improve genetic diagnosis and screening protocol of an at risk population.

The investigators hypothesize that siblings of patients with advanced neoplasm have an increased risk of both CRC and adenomas. The investigator aim to quantify this risk, and to identify other individual patient or neoplasm characteristics that may contribute to this increased risk. In addition, the investigator aim to determine molecular alteration profiles of colonic adenoma in siblings of patients with advanced neoplasm.

Investigator's preliminary data showed that the rate of advanced adenomas in controls (siblings of with normal colonoscopy) was 2%. Earlier studies have shown that the odds ratio of having colorectal neoplasms in close relatives of subjects with adenomas varies from 2.5 to 4.7. Using a conservative calculation, we assume that the prevalence of advanced adenomas in controls to be 3% and we estimate a 2.5-fold increased risk of advanced adenomas in siblings of individuals with advanced adenomas. Accordingly the recruitment of a minimum of 293 cases and 586 controls will be required to achieve 80% power to detect difference at a 5% significance level. For this project, investigators will aim to screen 300 siblings of patients with advanced adenomas and 600 matched controls.

ELIGIBILITY:
Inclusion Criteria:

* (case) Siblings (age > 40 and < 70) of individuals diagnosed with advanced neoplasm on screening colonoscopy. Advanced neoplasm is defined as adenomas ≥ 10mm size, >25% villous features, severe dysplasia or carcinoma-in-situ
* (control) Siblings of patients with negative findings on colonoscopy identified during the same study period, who are of the same age group as the studied cohort.

Exclusion Criteria:

* A family history compatible with that of Hereditary Non-polyposis Colon Cancer (HNPCC) based on the Amsterdam criteria [Table 3].
* Known Familial Adenomatous Polyposis (FAP) syndrome
* Patients and siblings with known inflammatory bowel disease
* Siblings that have undergone colonoscopy examinations in the past
* Severe cardio-pulmonary or other medical co-morbidities that preclude safe colonoscopic examination

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residence of Hong Kong siblings with colonoscopy done Siblings of Patients with Advanced Neoplasm (case) siblings of patients with normal colonoscopy (control)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-06-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adenoma and CRC | 30 days
  With informed consents, experienced colonoscopists will perform colonoscopy under intravenous sedation During colonoscopic examination, endoscopists are instructed to remove all raised lesions. The size, location and morphologic feature of each raised lesion will be recorded. The size is measured again an open biopsy forceps (6mm apart). To avoid observer bias, colonoscopists and pathologists will be blinded from patient's details regarding family history of CRC or advanced neoplasms. Our group performed the first screening study among average risk Hong Kong Chinese in the locality (28)

SECONDARY OUTCOMES:
Rate of advanced neoplasms depending on age of index case | 30 days
  same as primary outcome
Rate of advanced neoplasms depending on site of neoplasm | 30 days
  same as primary outcome
Differences in genetic profile between siblings of patients with advanced neoplasm and controls | 30 days
  same as primary outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Endoscopy Centre,Alice Ho Miu Ling Nethersole Hospital & Tai Po Hospital, Hong Kong, China
- Endocopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ng SC, Lau JY, Chan FK, Suen BY, Tse YK, Hui AJ, Leung-Ki EL, Ching JY, Chan AW, Wong MC, Ng SS, To KF, Wu JC, Sung JJ. Risk of Advanced Adenomas in Siblings of Individuals With Advanced Adenomas: A Cross-Sectional Study. Gastroenterology. 2016 Mar;150(3):608-16; quiz e16-7. doi: 10.1053/j.gastro.2015.11.003. Epub 2015 Nov 14. PMID 26584600